CLINICAL TRIAL: NCT01853878
Title: GSK2302032A Antigen-Specific Cancer Immunotherapeutic as Adjuvant Therapy in Patients With Non-Small Cell Lung Cancer
Brief Title: A Study to Demonstrate the Benefit of a New Kind of Anti-cancer Treatment [PReferentially Expressed Antigen of MElanoma (PRAME) Immunotherapy] for Patients With Non-Small Cell Lung Cancer (NSCLC), After Removal of Their Tumor
Acronym: PEARL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116389; 2012-002790-55 (EudraCT Number)
Record Dates: First submitted 2013-04-18; First posted 2013-05-15 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: Non-Small Cell Lung Cancer; Immunotherapy; Antigen-Specific
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- GSK2302032A Group (Experimental): The patients received 13 administrations GSK2302032A product, as per the following schedule: For the first five doses: 1 dose every 3 weeks. For the remaining 8 doses: 1 dose every 12 weeks.
  Interventions: Biological: Recombinant PRAME protein combined with the AS15 Adjuvant System GSK2302032A
- Placebo group (Placebo Comparator): The patients received 13 administrations of a placebo, as per the following schedule: For the first five doses: 1 dose every 3 weeks. For the remaining 8 doses: 1 dose every 12 weeks.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant PRAME protein combined with the AS15 Adjuvant System GSK2302032A — Intramuscular administration
  Arms: GSK2302032A Group
Biological: Placebo — Intramuscular administration
  Arms: Placebo group

SUMMARY:
The purpose of this study was to test a potential new kind of anti-cancer treatment, called PRAME immunotherapy in resected patients with lung cancer.

Based on scientific and medical relevance, the clinical study was ended on 24 August 2016. The participants were no longer enrolled in the study, the follow ups on subjects were stopped and the collection and analysis of samples for further research purposes was stopped.

After the stop to recruitment, the study was unblinded, as per the amended protocol, the study treatment was continued and completed with the subjects of the active treatment group who were willing to continue. Subjects in the placebo group were withdrawn.

There was no longer an active follow-up of patients after discontinuation or completion of the treatment. The study ended 30 days after the last dose was administered.

As a result, primary and secondary objectives were not assessed as planned. All clinical and safety data collected in the study were analysed descriptively. For each biological sample already collected in the scope of this study and not tested yet, testing was not performed by default, except if a scientific rationale remained relevant despite the premature termination of the study.

DETAILED DESCRIPTION:
During the treatment period, safety monitoring continued as initially foreseen. Reporting of post-study adverse events (AEs) and serious AEs (SAEs) continued as per protocol. In the best interest of the patient, no more biological samples for protocol research purposes (i.e. serum sampling for humoral immunity, whole blood sampling for pharmacogenetics) were taken.

ELIGIBILITY:
Inclusion Criteria:

* The patient has radically resected NSCLC
* The NSCLC is of pathological stage IA-T1b, IB, II or IIIA NSCLC The surgical technique for resection of the patient's tumor is anatomical, involving at least a segmentectomy The patient's tumor shows expression of PRAME.
* The patient is ≥ 18 years of age at the time of first consent.
* Written informed consent has been obtained from the patient prior to performance of any study-specific procedure.
* The patient is free of disease (no residual tumor, no loco-regional recurrence, no distant metastasis), as confirmed by a post- thoracic surgery contrast-enhanced computed tomography (CT scan) of the chest, upper abdomen and by a contrast-enhanced CT scan or Magnetic Resonance Imaging (MRI) of the brain. Other examinations should be performed as clinically indicated.
* Eastern Co-operative Oncology Group (ECOG) performance status of 0, 1 or 2 at the time of randomization
* Adequate bone-marrow reserve, adequate renal, hepatic and adrenal function as assessed by standard laboratory criteria
* If the patient is female, she must be of non-childbearing potential, i.e. have a current tubal ligation, hysterectomy, ovariectomy or be post-menopausal or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to administration of study product, have a negative pregnancy test and continue such precautions during all study treatment period and for 2 months after last treatment administration.
* Patients who the investigator believes can and will comply with the requirements of this protocol (e.g. return for active follow-up visits).

Exclusion Criteria:

* The patient is diagnosed with a concomitant malignancy and/or has a history of malignancy within the past five years or has had a malignancy that has been in complete remission for less than 5 years. Patients with effectively treated non - melanoma skin cancers or effectively treated carcinoma in situ of the cervix both of which in remission for less than 5 years will be eligible.
* The patient has received any anti-cancer specific treatment, including radiotherapy, immunotherapy, hormonal therapy, chemotherapy or neo-adjuvant chemotherapy, except for:

  * Administration of adjuvant platinum-based doublet chemotherapy for the treatment of the current NSCLC allowed between surgery and randomization.
  * Treatment of previous malignancies as allowed by the protocol.
* The patient has been diagnosed with a Potential Immune-Mediated Disease (pIMD). Patients with vitiligo are not excluded from the study.
* The patient has a history of confirmed adrenal dysfunction.
* The patient requires concomitant treatment with any immunosuppressive agent, or with systemic corticosteroids prescribed for chronic treatment (more than 7 consecutive days).
* The patient needs chronic long term oxygen therapy (LTOT). The patient has medically uncontrolled congestive heart failure or hypertension, unstable heart disease or uncontrolled arrhythmia at the time of randomization.
* The patient has an uncontrolled bleeding disorder.
* The patient has undergone splenectomy.
* The patient is known to be Human Immunodeficiency Virus (HIV)-positive.
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the trial procedures.
* The patient has other concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* The patient has a history of allergic disease or reactions likely to be exacerbated by any component of the study investigational product.
* The patient has received any investigational or non-registered product within the 30 days preceding randomization, or planned use during the study period.
* For female patients: the patient is pregnant or lactating or is planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2013-06-12 (Actual); Primary Completion 2016-08-24 (Actual); Study Completion 2016-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (37):
- United States (8):
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Paterson, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Seattle, Washington
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (4):
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
- Germany (10):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Immenhausen, Hesse
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Moers, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Japan (3):
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Shizuoka
- Poland (2):
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Zakopane
- Russia (2):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Saint Petersburg
- GSK Investigational Site, Seoul, South Korea
- United Kingdom (5):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below).
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 116389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116389 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: On 18 July 2014, the recruitment was stopped and the study was un-blinded. The study continued only with patients from the active treatment group who decided to stay in the study, however objective and outcomes were not assessed as planned.
Pre-assignment Details: Among 137 enrolled patients, 4 patients didn't receive any study product dose and hence they were not taken into account for study start.
Period: Overall Study
Arm/Group | GSK2302032A Group | Placebo Group
Started | 86 | 47
Completed | 23 | 3
Not Completed | 63 | 44
Not completed — Recurrence | 2 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Migrated/moved from the study area | 1 | 0
Not completed — Other | 55 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2302032A Group | Placebo Group | Total
Number analyzed (Participants) | 86 | 47 | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (8.68) | 62.7 (9.28) | 63.86 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 13 | 39
  Male | 60 | 34 | 94
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Occurrence of Any Recurrence of Disease
Description: Time to occurrence of any recurrence of disease was expressed in terms of rate: Person-year rate in each group = number of patients reporting at least one recurrence of disease (n)/ sum of follow-up period expressed in years (T[year)]) As a consequence of the decision to stop the PRAME-AS15-NSC-002 (ADJ) study, not all data were available for a full analysis. The median follow-up time was 10.3 months in the GSK2302032A group and 5.7 months in the Placebo group. Considering that two Phase III studies with recMAGE-A3 + AS15 failed to demonstrate clinical efficacy of the MAGE-A3 antigen specific cancer immunotherapeutic, GSK decided to stop the development of all recombinant protein based cancer vaccines and to stop recruitment in all the ongoing clinical studies.
Time Frame: During the entire study (From Week 1 to Week 112)
Population: The analysis was performed on the Total Treated population that included all the subjects who had received at least one dose of the study product.
Measure: Number; unit: person-year rate
Arm/Group | GSK2302032A Group | Placebo Group
Number analyzed (Participants) | 86 | 47
person-year rate | 0.217 | 0.067
Statistical Analysis 1: Comparison: GSK2302032A Group vs Placebo Group; Estimates of Hazard Ratio (HR) and their 95% Confidence Interval (CI) were obtained by Cox regression modelling.The Likelihood ratio test was used to compare the groups. The Cox proportional hazard regression was stratified by previous treatment [Chemotherapy (CT) vs. no-CT] and disease stage; Test type: Equivalence — P-value of the Wald test from a Cox regression model to test H0 = { HR=1} (Y = Time to Event); p = 0.1422, Regression, Cox; Hazard Ratio (HR) = 4.592, 95% CI 2-sided [0.600 to 35.167]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the interval from randomization to the date of death, irrespective of the cause of death; patients still alive were censored at the last visit they are known to be alive. Considering that two Phase III studies with recMAGE-A3 + AS15 failed to demonstrate clinical efficacy of the MAGE-A3 antigen specific cancer immunotherapeutic, GSK decided to stop the development of all recombinant protein based cancer vaccines and to stop recruitment in all the ongoing clinical studies. Therefore, based on scientific and medical relevance, the decision was made to stop patient enrollment in the PRAME-AS15-NSC-002 (ADJ) clinical study and to stop follow-up visits, further sample collection for research purposes and the analysis of samples for research purposes. In consequence, the primary and secondary outcomes were not analysed as planned and clinical data for this outcome was not collected.
Time Frame: During the entire study (From Week 1 to Week 112)
Population: Overall survival data was not collected.
Arm/Group | GSK2302032A Group | Placebo Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Lung-cancer-specific Survival
Description: Lung-cancer specific survival was defined as defined as the interval from randomization to the date of death due to lung cancer; deaths due to other or unknown causes were censored at the date of death. Considering that two Phase III studies with recMAGE-A3 + AS15 failed to demonstrate clinical efficacy of the MAGE-A3 antigen specific cancer immunotherapeutic, GSK decided to stop the development of all recombinant protein based cancer vaccines and to stop recruitment in all the ongoing clinical studies. Therefore, based on scientific and medical relevance, the decision was made to stop patient enrollment in the PRAME-AS15-NSC-002 (ADJ) clinical study and to stop follow-up visits, further sample collection for research purposes and the analysis of samples for research purposes. In consequence, the primary and secondary outcomes were not analysed as planned and clinical data for this outcome was not collected.
Time Frame: During the entire study (From Week 1 to Week 112)
Population: Lung-cancer specific survival data was not collected.
Arm/Group | GSK2302032A Group | Placebo Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Disease-free Specific Survival (DFSS)
Description: DFSS was defined as the interval from randomization to the date of first recurrence of disease or date of death due to lung cancer, whichever occurs first. Patients without recurrence or death due to lung cancer were censored at the date of last assessment. Considering that two Phase III studies with recMAGE-A3 + AS15 failed to demonstrate clinical efficacy of the MAGE-A3 antigen specific cancer immunotherapeutic, GSK decided to stop the development of all recombinant protein based cancer vaccines and to stop recruitment in all the ongoing clinical studies. Therefore, based on scientific and medical relevance, the decision was made to stop patient enrollment in the PRAME-AS15-NSC-002 (ADJ) clinical study and to stop follow-up visits, further sample collection for research purposes and the analysis of samples for research purposes. In consequence, the primary and secondary outcomes were not analysed as planned and clinical data for this outcome was not collected.
Time Frame: During the entire study (From Week 1 to Week 112)
Population: Disease free-specific survival data was not collected.
Arm/Group | GSK2302032A Group | Placebo Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: DFS (Disease-free Survival) at 2, 3, 4 and 5 Years After Randomization
Description: Defined as the time from randomization to either the date of first recurrence of the disease or the date of death (whatever the cause), whichever occurred first. The 5-year active follow-up period planned in the initial study protocol was cancelled per Protocol Amendment 2, hence this analysis was not performed.
Time Frame: During the entire follow-up period (From year 2 to Year 5)
Population: The 5-Year Follow-Up Disease Free Survival data were not collected.
Arm/Group | GSK2302032A Group | Placebo Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs covered any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 31-day (Days 0-30) post-vaccine administration period
Population: This analysis was performed on the Total Treated population, which included all the patients who had received at least one dose of the study product.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302032A Group | Placebo Group
Number analyzed (Participants) | 86 | 47
Participants | 78 | 21

7. Secondary Outcome: Anti-PRAME Antibody Concentrations
Description: Considering that two Phase III studies with recMAGE-A3 + AS15 failed to demonstrate clinical efficacy of the MAGE-A3 antigen specific cancer immunotherapeutic, GSK decided to stop the development of all recombinant protein based cancer vaccines and to stop recruitment in all the ongoing clinical studies. Therefore, based on scientific and medical relevance, the decision was made to stop patient enrollment in the PRAME-AS15-NSC-002 (ADJ) clinical study and to stop follow-up visits, further sample collection for research purposes and the analysis of samples for research purposes. In consequence, the primary and secondary outcomes were not analysed as planned and clinical data for this outcome was not collected.
Time Frame: At each defined time point from Week 0 till Concluding Visit (Week 112)
Population: Anti-PRAME antibody data was not collected.
Arm/Group | GSK2302032A Group | Placebo Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Subjects With Any Abnormal Hematological and Biochemical Parameters
Description: Hematological and biochemical parameters assessed were tabulated by maximum grade versus baseline, by CTCAE = Common Terminology Criteria for Adverse Events version 4.0 (Grade 1= mild; Grade 2= moderate; Grade 3= severe; Grade 4= life-threatening; Grade 5 = death; Grade Unknown) and by the type of abnormality (e.g. increased, decreased, prolonged, etc.). Some parameters (e.g. Anemia) already comprise within their definition the type of abnormality presented.
Time Frame: During the entire study period (From Week 1 to Week 112)
Population: This analysis was performed on the Total Treated population, which included all the patients who had received at least one dose of the study product and for whom blood results were available for the respective parameter assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302032A Group | Placebo Group
Number analyzed (Participants) | 86 | 47
Participants
  Activated partial thromboplastin time prolonged: number analyzed (Participants) | 28 | 10
  Activated partial thromboplastin time prolonged: Grade 1 | 26 | 8
  Activated partial thromboplastin time prolonged: Grade 2 | 1 | 0
  Activated partial thromboplastin time prolonged: Grade 3 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 4 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 5 | 0 | 0
  Activated partial thromboplastin time prolonged: Unknown | 1 | 2
  Alanine aminotransferase increased: number analyzed (Participants) | 18 | 7
  Alanine aminotransferase increased: Grade 1 | 17 | 6
  Alanine aminotransferase increased: Grade 2 | 1 | 0
  Alanine aminotransferase increased: Grade 3 | 0 | 0
  Alanine aminotransferase increased: Grade 4 | 0 | 0
  Alanine aminotransferase increased: Grade 5 | 0 | 0
  Alanine aminotransferase increased: Unknown | 0 | 1
  Alkaline Phosphatase increased: number analyzed (Participants) | 17 | 6
  Alkaline Phosphatase increased: Grade 1 | 17 | 5
  Alkaline Phosphatase increased: Grade 2 | 0 | 0
  Alkaline Phosphatase increased: Grade 3 | 0 | 0
  Alkaline Phosphatase increased: Grade 4 | 0 | 0
  Alkaline Phosphatase increased: Grade 5 | 0 | 0
  Alkaline Phosphatase increased: Unknown | 0 | 1
  Anemia: number analyzed (Participants) | 37 | 20
  Anemia: Grade 1 | 36 | 17
  Anemia: Grade 2 | 0 | 2
  Anemia: Grade 3 | 0 | 0
  Anemia: Grade 4 | 0 | 0
  Anemia: Grade 5 | 0 | 0
  Anemia: Unknown | 1 | 1
  Aspartate aminotransferase increased: number analyzed (Participants) | 15 | 6
  Aspartate aminotransferase increased: Grade 1 | 15 | 5
  Aspartate aminotransferase increased: Grade 2 | 0 | 0
  Aspartate aminotransferase increased: Grade 3 | 0 | 0
  Aspartate aminotransferase increased: Grade 4 | 0 | 0
  Aspartate aminotransferase increased: Grade 5 | 0 | 0
  Aspartate aminotransferase increased: Unknown | 0 | 1
  Blood bilirubin increased: number analyzed (Participants) | 8 | 4
  Blood bilirubin increased: Grade 1 | 7 | 2
  Blood bilirubin increased: Grade 2 | 1 | 1
  Blood bilirubin increased: Grade 3 | 0 | 0
  Blood bilirubin increased: Grade 4 | 0 | 0
  Blood bilirubin increased: Grade 5 | 0 | 0
  Blood bilirubin increased: Unknown | 0 | 1
  Creatinine increased: number analyzed (Participants) | 18 | 8
  Creatinine increased: Grade 1 | 15 | 7
  Creatinine increased: Grade 2 | 3 | 0
  Creatinine increased: Grade 3 | 0 | 0
  Creatinine increased: Grade 4 | 0 | 0
  Creatinine increased: Grade 5 | 0 | 0
  Creatinine increased: Unknown | 0 | 1
  Gamma-glutamyl transferase increased: number analyzed (Participants) | 23 | 14
  Gamma-glutamyl transferase increased: Grade 1 | 14 | 11
  Gamma-glutamyl transferase increased: Grade 2 | 7 | 1
  Gamma-glutamyl transferase increased: Grade 3 | 2 | 0
  Gamma-glutamyl transferase increased: Grade 4 | 0 | 0
  Gamma-glutamyl transferase increased: Grade 5 | 0 | 0
  Gamma-glutamyl transferase increased: Unknown | 0 | 2
  Hemoglobin increased: number analyzed (Participants) | 6 | 2
  Hemoglobin increased: Grade 1 | 5 | 1
  Hemoglobin increased: Grade 2 | 1 | 0
  Hemoglobin increased: Grade 3 | 0 | 0
  Hemoglobin increased: Grade 4 | 0 | 0
  Hemoglobin increased: Grade 5 | 0 | 0
  Hemoglobin increased: Unknown | 0 | 1
  Hyperkalemia: number analyzed (Participants) | 27 | 14
  Hyperkalemia: Grade 1 | 22 | 12
  Hyperkalemia: Grade 2 | 4 | 1
  Hyperkalemia: Grade 3 | 1 | 0
  Hyperkalemia: Grade 4 | 0 | 0
  Hyperkalemia: Grade 5 | 0 | 0
  Hyperkalemia: Unknown | 0 | 1
  Hypernatremia: number analyzed (Participants) | 17 | 8
  Hypernatremia: Grade 1 | 13 | 6
  Hypernatremia: Grade 2 | 4 | 1
  Hypernatremia: Grade 3 | 0 | 0
  Hypernatremia: Grade 4 | 0 | 0
  Hypernatremia: Grade 5 | 0 | 0
  Hypernatremia: Unknown | 0 | 1
  Hypoalbuminemia: number analyzed (Participants) | 21 | 12
  Hypoalbuminemia: Grade 1 | 18 | 10
  Hypoalbuminemia: Grade 2 | 3 | 0
  Hypoalbuminemia: Grade 3 | 0 | 0
  Hypoalbuminemia: Grade 4 | 0 | 0
  Hypoalbuminemia: Grade 5 | 0 | 0
  Hypoalbuminemia: Unknown | 0 | 2
  Hypokalemia: number analyzed (Participants) | 3 | 2
  Hypokalemia: Grade 1 | 3 | 1
  Hypokalemia: Grade 2 | 0 | 0
  Hypokalemia: Grade 3 | 0 | 0
  Hypokalemia: Grade 4 | 0 | 0
  Hypokalemia: Grade 5 | 0 | 0
  Hypokalemia: Unknown | 0 | 1
  Hyponatremia: number analyzed (Participants) | 11 | 7
  Hyponatremia: Grade 1 | 10 | 6
  Hyponatremia: Grade 2 | 0 | 0
  Hyponatremia: Grade 3 | 1 | 0
  Hyponatremia: Grade 4 | 0 | 0
  Hyponatremia: Grade 5 | 0 | 0
  Hyponatremia: Unknown | 0 | 1
  Lymphocyte count decreased: number analyzed (Participants) | 24 | 11
  Lymphocyte count decreased: Grade 1 | 19 | 8
  Lymphocyte count decreased: Grade 2 | 3 | 2
  Lymphocyte count decreased: Grade 3 | 2 | 0
  Lymphocyte count decreased: Grade 4 | 0 | 0
  Lymphocyte count decreased: Grade 5 | 0 | 0
  Lymphocyte count decreased: Unknown | 0 | 1
  Lymphocyte count increased: number analyzed (Participants) | 2 | 1
  Lymphocyte count increased: Grade 1 | 0 | 0
  Lymphocyte count increased: Grade 2 | 2 | 0
  Lymphocyte count increased: Grade 3 | 0 | 0
  Lymphocyte count increased: Grade 4 | 0 | 0
  Lymphocyte count increased: Grade 5 | 0 | 0
  Lymphocyte count increased: Unknown | 0 | 1
  Neutrophil count decreased: number analyzed (Participants) | 13 | 9
  Neutrophil count decreased: Grade 1 | 9 | 7
  Neutrophil count decreased: Grade 2 | 4 | 1
  Neutrophil count decreased: Grade 3 | 0 | 0
  Neutrophil count decreased: Grade 4 | 0 | 0
  Neutrophil count decreased: Grade 5 | 0 | 0
  Neutrophil count decreased: Unknown | 0 | 1
  Platelet count decreased: number analyzed (Participants) | 7 | 2
  Platelet count decreased: Grade 1 | 6 | 1
  Platelet count decreased: Grade 2 | 1 | 0
  Platelet count decreased: Grade 3 | 0 | 0
  Platelet count decreased: Grade 4 | 0 | 0
  Platelet count decreased: Grade 5 | 0 | 0
  Platelet count decreased: Unknown | 0 | 1
  White blood cell decreased: number analyzed (Participants) | 8 | 5
  White blood cell decreased: Grade 1 | 7 | 4
  White blood cell decreased: Grade 2 | 1 | 0
  White blood cell decreased: Grade 3 | 0 | 0
  White blood cell decreased: Grade 4 | 0 | 0
  White blood cell decreased: Grade 5 | 0 | 0
  White blood cell decreased: Unknown | 0 | 1

9. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed included medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. An event that was part of the natural course of the disease under study (i.e., disease progression, recurrence) was captured in the study as an efficacy measure; therefore it did not need to be reported as an SAE.
Time Frame: During the entire study (From Week 1 to Week 112)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302032A Group | Placebo Group
Number analyzed (Participants) | 86 | 47
Participants | 14 | 0

10. Secondary Outcome: Number of Subjects With Any Adverse Events (AEs) by Intensity Grade.
Description: Grading was done as per the Common Terminology Criteria for Adverse Events (CTCAE) of the U.S. National Cancer Institute, version 4.0. The intensity grades assessed were: 1, 2, 3, 4, 5 and Unknown.
Time Frame: From Week 0 to Week 112
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302032A Group | Placebo Group
Number analyzed (Participants) | 86 | 47
Participants
  Any Grade 1 AEs | 35 | 17
  Any Grade 2 AEs | 29 | 8
  Any Grade 3 AEs | 15 | 2
  Any Grade 4 AEs | 3 | 0
  Any Grade 5 AEs | 1 | 0
  Any Grade Unknown AEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events: within the 31-day (Days 0-30) period following study treatment administration. Serious adverse events (SAEs): throughout the study (i.e. up to Week 112).
Description: An event that was part of the natural course of the disease under study (i.e., disease progression, recurrence) was captured in the study as an efficacy measure; therefore it did not need to be reported as an SAE.
Arm/Group | GSK2302032A Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 1/86 | 0/47
Serious Adverse Events (participants affected / at risk) | 14/86 | 0/47
Other Adverse Events (participants affected / at risk) | 78/86 | 21/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2302032A Group (N=86) | Placebo Group (N=47)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Hemorrhagic pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.13% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2302032A Group (N=86) | Placebo Group (N=47)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (11) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (7) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 6 (21) | 1 (1)
Fatigue (General disorders) | 14 (35) | 7 (10)
Influenza like illness (General disorders) | 16 (59) | 2 (3)
Injection site erythema (General disorders) | 18 (31) | 1 (1)
Injection site pain (General disorders) | 49 (175) | 1 (2)
Injection site reaction (General disorders) | 12 (42) | 0 (0)
Injection site swelling (General disorders) | 6 (16) | 0 (0)
Malaise (General disorders) | 5 (15) | 0 (0)
Pain (General disorders) | 4 (8) | 1 (1)
Pyrexia (General disorders) | 35 (132) | 1 (5)
Bronchitis (Infections and infestations) | 1 (2) | 2 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 0 (0)
Headache (Nervous system disorders) | 6 (11) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 3 (3)

LIMITATIONS AND CAVEATS:
As of 18 July 2014, the recruitment was stopped and the study was unblinded. For patients randomized to the placebo group, no further protocol visits were to be performed except for the concluding visit and no further doses were to be administered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.